CLINICAL TRIAL: NCT00727064
Title: A Randomized, Open-Label, Two-Period, Parallel Group, Crossover Study to Evaluate the Pharmacokinetics of Venlafaxine Extended-Release and DVS SR in Healthy Subjects Who Are Extensive or Poor Cytochrome P450 2D6 Substrate Metabolizers
Brief Title: Study Evaluating the Pharmacokinetics of Venlafaxine Extended-Release (ER) and Desvenlafaxine Succinate Sustained-Release (DVS SR) 50 mg in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 3151A1-4414
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Results first posted 2010-04-19 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Healthy
Keywords: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DVS/VEN (Active Comparator)
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release (DVS SR); Drug: Venlafaxine Extended Release (VEN ER)
- VEN/DVS (Active Comparator)
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release (DVS SR); Drug: Venlafaxine Extended Release (VEN ER)

INTERVENTIONS:
Drug: Desvenlafaxine Succinate Sustained-Release (DVS SR)
Drug: Venlafaxine Extended Release (VEN ER)

SUMMARY:
The purpose of this study is to determine if the relative difference in Pharmacokinetics (PK) between extensive metabolizers (EMs) and poor metabolizers (PMs) is the same with desvenlafaxine SR and venlafaxine ER when a single dose is administered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 18 to 55 years. Healthy as determined by the investigator on the basis of medical history and physical examination, laboratory test results, vital signs, and 12-lead electrocardiogram (ECG).
* History of being a nonsmoker for at least 1 year.
* Subjects have to be either extensive CYP2D6 metabolizers with a normal complement of 1 or 2 fully active enzyme gene alleles or poor CYP2D6 metabolizers (lack of active enzyme gene alleles) via genetic testing of a blood sample.

Exclusion Criteria:

* Presence or history of any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease or any severe conditions of the ears, eyes or throat (such as glaucoma or increased intraocular pressure).
* Known or suspected alcohol abuse or consumption of more than 2 standard units per day (a standard unit equals 12 ounces of beer, 1½ ounces of 80-proof alcohol, or 6 ounces of wine) within the past 6 months.
* Known or suspected current abuse of prohibited drugs or other substances. Use of any hormonal therapy within 30 days before study day -1 until the end of the partial inpatient confinement period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Clinical Research Institute, Wichita, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in the United States from June 2008 to August 2008.
Pre-assignment Details: Participants were screened for cytochrome P450 2D6 (CYP2D6) genotype to identify 7 "extensive metabolizers" and 7 "poor metabolizers" (inclusion criteria). Eligible participants were then randomly assigned to a sequence group.
Groups:
- Sequence Group A: Day 1: single 50mg oral dose of Desvenlafaxine Succinate Sustained Release (DVS SR) in a fasting state. Days 1-6: 120 hours of PK sampling. Days 7-10: Wash out period. Day 11: single 75mg oral dose of Venlafaxine ER (VEN ER) in a fasting state. Day 11-16: 120 hours of PK sampling.
- Sequence Group B: Day 1: single 75mg oral dose of Venlafaxine Extended Release (VEN ER) in a fasting state. Days 1-6: 120 hours of PK sampling. Days 7-10: Wash out period. Day 11: single 50mg oral dose of Desvenlafaxine Succinate Sustained Release (DVS SR) in a fasting state. Day 11-16: 120 hours of PK sampling.
Period: Overall Study
Arm/Group | Sequence Group A | Sequence Group B
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence Group A | Sequence Group B | Total
Number analyzed (Participants) | 7 | 7 | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 30.14 (10.37) | 28.29 (8.90) | 29.21 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax) of Venlafaxine After Single Dose of Venlafaxine Extended-release (VEN ER) by Metabolizer Status
Description: Cmax is a measure of drug metabolism and presented as least squares geometric mean with 90% Confidence Interval. Variations in drug metabolism among individuals can be due to differences in genetic expression (phenotype) of Cytochrome P450 (CYP450) enzymes. Enzyme CYP2D6 has 4 metabolizer phenotypes: poor (PM), intermediate (IM), extensive (EM), and ultrarapid (UM) metabolizers.
Time Frame: single dose
Population: All participants from sequence groups A and B who received a single dose of venlafaxine ER.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL (90% CI)
Groups:
- Extensive Metabolizers (EM): Identified as EM from CYP2D6 testing at screening
- Poor Metabolizers (PM): Identified as PM from CYP2D6 testing at screening
Arm/Group | Extensive Metabolizers (EM) | Poor Metabolizers (PM)
Number analyzed (Participants) | 7 | 7
ng/mL (90% CI) | 26.16 (17.70) [20.01 to 34.19] | 77.46 (32.36) [59.25 to 101.25]
Statistical Analysis 1: Comparison: Extensive Metabolizers (EM) vs Poor Metabolizers (PM); Test type: Superiority or Other; p < 0.001, ANOVA; PM compared to EM using least squares geometric means. Analysis of variance with phenotype and sequence as factors

2. Primary Outcome: Area Under the Concentration-time Curve (AUC) of Venlafaxine After Single Dose of VEN ER by Metabolizer Status
Description: AUC is drug level over time and measures drug metabolism. Variations in drug metabolism among individuals can be due to differences in genetic expression (phenotype) of Cytochrome P450 (CYP450) enzymes. Enzyme CYP2D6 has 4 metabolizer phenotypes: poor (PM), intermediate (IM), extensive (EM), ultrarapid (UM) metabolizers.
Time Frame: single dose
Population: All participants from sequence groups A and B who received a single dose of venlafaxine ER.
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL (90% CI)
Arm/Group | Extensive Metabolizers (EM) | Poor Metabolizers (PM)
Number analyzed (Participants) | 7 | 7
ng*h/mL (90% CI) | 389.68 (462.45) [247.02 to 614.72] | 2328.41 (3460.47) [1475.99 to 3673.13]
Statistical Analysis 1: Comparison: Extensive Metabolizers (EM) vs Poor Metabolizers (PM); Test type: Superiority or Other; p < 0.001, ANOVA; PM compared to EM using least squares geometric means. Analysis of variance with phenotype and sequence as factors

3. Primary Outcome: Maximum Concentration (Cmax) of Desvenlafaxine After Single Dose of VEN ER by Metabolizer Status
Description: Cmax is a measure of drug metabolism. Variations in drug metabolism among individuals can be due to differences in genetic expression (phenotype) of Cytochrome P450 (CYP450) enzymes. Enzyme CYP2D6 has 4 metabolizer phenotypes: poor (PM), intermediate (IM), extensive (EM), and ultrarapid (UM) metabolizers.
Time Frame: single dose
Population: All participants from sequence groups A and B who received a single dose of venlafaxine ER.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL (90% CI)
Arm/Group | Extensive Metabolizers (EM) | Poor Metabolizers (PM)
Number analyzed (Participants) | 7 | 7
ng/mL (90% CI) | 95.63 (27.40) [51.77 to 176.68] | 15.73 (20.27) [8.51 to 29.06]
Statistical Analysis 1: Comparison: Extensive Metabolizers (EM) vs Poor Metabolizers (PM); Test type: Superiority or Other; p = 0.004, ANOVA; PM compared to EM using least squares geometric means. Analysis of variance with phenotype and sequence as factors

4. Primary Outcome: Area Under the Concentration-time Curve (AUC) of Desvenlafaxine After Single Dose of VEN ER by Metabolizer Status
Description: as for outcome 2
Time Frame: single dose
Population: All participants from sequence groups A and B who received a single dose of venlafaxine ER.
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL (90% CI)
Arm/Group | Extensive Metabolizers (EM) | Poor Metabolizers (PM)
Number analyzed (Participants) | 7 | 7
ng*h/mL (90% CI) | 2703.50 (540.96) [1191.90 to 6132.19] | 436.14 (442.86) [192.28 to 989.26]
Statistical Analysis 1: Comparison: Extensive Metabolizers (EM) vs Poor Metabolizers (PM); Test type: Superiority or Other; p = 0.018, ANOVA; PM compared to EM using least squares geometric means. Analysis of variance with phenotype and sequence as factors

5. Primary Outcome: Maximum Concentration (Cmax) of Desvenlafaxine After Single Dose of Desvenlafaxine Succinate Sustained-Release (DVS SR) by Metabolizer Status
Description: Cmax is a measure of drug metabolism and is presented as least squares geometric mean with 90% Confidence Interval.Variations in drug metabolism among individuals can be due to differences in genetic expression (phenotype) of Cytochrome P450 (CYP450) enzymes. Enzyme CYP2D6 has 4 metabolizer phenotypes: poor (PM), intermediate (IM), extensive (EM), and ultrarapid (UM) metabolizers.
Time Frame: single dose
Population: All participants from sequence groups A and B who received a single dose of venlafaxine ER.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL (90% CI)
Arm/Group | Extensive Metabolizers (EM) | Poor Metabolizers (PM)
Number analyzed (Participants) | 7 | 7
ng/mL (90% CI) | 102.22 (15.35) [83.52 to 125.12] | 125.32 (28.34) [101.80 to 154.28]
Statistical Analysis 1: Comparison: Extensive Metabolizers (EM) vs Poor Metabolizers (PM); Test type: Superiority or Other; p = 0.081, ANOVA; PM compared to EM using least squares geometric means. Analysis of variance with phenotype and sequence as factors

6. Primary Outcome: Area Under the Concentration-time Curve (AUC) of Desvenlafaxine After Single Dose of DVS SR by Metabolizer Status
Description: as for outcome 2
Time Frame: single dose
Population: All participants from sequence groups A and B who received a single dose of venlafaxine ER.
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL (90% CI)
Arm/Group | Extensive Metabolizers (EM) | Poor Metabolizers (PM)
Number analyzed (Participants) | 7 | 7
ng*h/mL (90% CI) | 2701.79 (414.79) [2024.74 to 3605.25] | 3111.25 (1050.76) [2316.01 to 4179.55]
Statistical Analysis 1: Comparison: Extensive Metabolizers (EM) vs Poor Metabolizers (PM); Test type: Superiority or Other; p = 0.427, ANOVA; PM compared to EM using least squares geometric means. Analysis of variance with phenotype and sequence as factors

ADVERSE EVENTS:
Groups:
- Desvenlafaxine Succinate Sustained-Release (DVS SR): SAE or AE reported on DVS SR regardless of which arm or period of trial.
- Venlafaxine Extended Release (VEN ER): SAE or AE reported on VEN ER regardless of which arm or period of trial.
Arm/Group | Desvenlafaxine Succinate Sustained-Release (DVS SR) | Venlafaxine Extended Release (VEN ER)
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 2 | 4
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Desvenlafaxine Succinate Sustained-Release (DVS SR) | Venlafaxine Extended Release (VEN ER)
Nausea (Gastrointestinal disorders) | 1/7 | 1/7
Headache (Nervous system disorders) | 0/7 | 2/7
Syncope vasovagal (Nervous system disorders) | 0/7 | 1/7
Insomina (Psychiatric disorders) | 1/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.